CLINICAL TRIAL: NCT00998283
Title: A Randomized, Double-Blind, Placebo-Controlled, Escalating Single-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of HM10460A (HNK460) When Administered Subcutaneously to Healthy Adult Korean Subjects
Brief Title: Assess the Safety, Tolerability, and Pharmacokinetic (PK) Characteristics of HM10460A (HNK460) in Healthy Adult Korean Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-HM10460A-102
Record Dates: First submitted 2009-10-18; First posted 2009-10-20 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
MeSH Terms: interventions — eflapegrastim

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Experimental): Administration of HM10460A 5μg/kg or Placebo
  Interventions: Drug: HM10460A 5μg/kg; Drug: Placebo
- Cohort 2 (Experimental): Administration of HM10460A 15μg/kg or placebo
  Interventions: Drug: HM10460A 15μg/kg; Drug: Placebo
- Cohort 3 (Experimental): Administration of HM10460A 45μg/kg or placebo
  Interventions: Drug: HM10460A 45μg/kg; Drug: Placebo
- Cohort 4 (Experimental): Administration of HM10460A 135μg/kg or placebo
  Interventions: Drug: HM10460A 135μg/kg; Drug: Placebo
- Cohort 5 (Experimental): Administration of HM10460A 350μg/kg or placebo
  Interventions: Drug: HM10460A 350μg/kg; Drug: Placebo

INTERVENTIONS:
Drug: HM10460A 5μg/kg — Subcutaneously administrate at 0 hour on Day 1
  Arms: Cohort 1
Drug: HM10460A 15μg/kg — Subcutaneously administrate at 0 hour on Day 1
  Arms: Cohort 2
Drug: HM10460A 45μg/kg — Subcutaneously administrate at 0 hour on Day 1
  Arms: Cohort 3
Drug: HM10460A 135μg/kg — Subcutaneously administrate at 0 hour on Day 1
  Arms: Cohort 4
Drug: HM10460A 350μg/kg — Subcutaneously administrate at 0 hour on Day 1
  Arms: Cohort 5
Drug: Placebo — Subcutaneously administrate at 0 hour on Day 1

SUMMARY:
* Study Design

  * Randomized, Double-blind, Placebo-controlled, escalating single-dose design.
  * Five ascending dose cohorts.
  * In each cohort, subjects will be randomized to receive a single dose of HM10460A or placebo (negative control)
* Objectives

  * The primary objective of the study is to assess the safety and tolerability of single escalating subcutaneous doses of HM10460A in healthy adult Korean Subjects

DETAILED DESCRIPTION:
The secondary objectives of the study are as follows:

* to assess the pharmacokinetics (PK) of a single subcutaneous dose of HM10460A.
* to assess the relationship between the serum concentration of HM10460A and absolute neutrophil count (ANC).
* to assess the relationship between the serum concentration of HM10460A and CD34+ cell counts in the blood.
* to assess the immunogenicity (HM10460A, native G-CSF antibody,neutralizing antibodies) of a single subcutaneous dose of HM10460A.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult Korean male and/or females, 20 - 45 years of age(inclusive).
* BMI of 18 - 27kg/m2.
* Medically healthy with no clinically significant screening results.
* The following results in laboratory test
* Absolute neutrophil count (ANC) : 2000 ~ 7500/mm3
* Non-smokers or subjects who smoke less than 10 cigarettes/day
* After a confirmed menstrual period, females of childbearing potential must be either sexually inactive (abstinent) for 14 days prior to screening and agree to remain so throughout the study, or have been using a highly effective method of birth control, such as the following examples:

  * intra-uterine device in place for at least 3 months prior to Day 1;
  * stable hormonal contraceptive for at least 3 months prior to Day 1 through completion of study;
  * surgical sterilization (vasectomy) of partner at least 6 months prior to Day 1.
* Females of non-childbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to Day 1:

  * bilateral tubal ligation;
  * hysterectomy;
  * hysterectomy with unilateral or bilateral oophorectomy;
  * bilateral oophorectomy.

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
* Positive urine drug/alcohol testing at screening or check-in.
* Positive testing for HIV, HBsAg, or HCV antibodies.
* Active infection
* Positive testing for palpable spleen at screening or check-in.
* The following results in laboratory test:

  * WBC > 10.0 x 10^3/mm3
  * Hb < 13g/dL
  * Platelet < 150 x 10^3/mm3
  * AST/ALT > 50 IU/L
* History or presence of alcoholism or drug abuse within 2 years prior to Day 1.
* History of G-CSF-related product use (i.e., pegfilgrastim, filgrastim).
* History of anaphylactic reaction to medicine or environmental exposures.
* Use of any prescription medication (with the exception of hormonal contraceptives for females) or receipt of any blood products within 14 days prior to Day 1.
* Use of any over-the-counter medication, including herbal products, within 7 days prior to the Day 1. Up to 2 grams per day of acetaminophen is allowed at the discretion of the Investigator.
* Blood donation or significant blood loss within 56 days prior to Day 1.
* Plasma donation within 7 days prior to Day 1.
* Participation in another clinical trial (receipt of last investigational medication) within 30 days prior to Day 1.
* Females who are pregnant or lactating.
* Subjects who are unlikely to comply with the protocol requirements, instructions and study related restrictions; e.g., uncooperative attitude, inability to return for follow-up visits and improbability of completing the clinical study.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety data, including physical examinations (to include injection site reactions and splenic evaluations), laboratory evaluations, ECGs, vital signs, and adverse effects (AEs) | Time point of collection, where appropriate
Samples for immunogenicity | Time point of collection, where appropriate

SECONDARY OUTCOMES:
Serum PK parameters/Urine PK parameters | Serum : pre-dose, 0.25, 05, 0.75, 1,2,3,4,6,8,12,16,24,36,48,72,96,120,144 (hr)// Urine : 0-6, 6-12, 12-24, 24-36, 36,48(hr)
Calculation of the ANC (Absolute Neutrophil count) & CD34+ cell. | Pre-dose, 24 and 48 hours post-dose, on return Days 4,5,6,7,11,15 and 22

CONTACTS AND LOCATIONS:
Overall Officials: Hanmi Clinical, Principal Investigator — Seoul
Locations (1):
- Seoul, South Korea